CLINICAL TRIAL: NCT06355089
Title: Intestinal Microbiota: Immunity, Recovery and Metabolic Health
Acronym: VAR-MIKRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Government Body Funding (Unknown)
Responsible Party: Principal Investigator, Kirsi Laitinen, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: VAR-MIKRO
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Nutrition; Probiotics; Whey protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo milk product (Placebo Comparator): Use of low protein milk product
  Interventions: Dietary Supplement: Placebo Comparator
- Whey protein hydrolysate milk product (Active Comparator): Use of milk product with whey protein hydrolysate
  Interventions: Dietary Supplement: Whey protein hydrolysate milk product
- Postbiotic and whey protein hydrolysate milk product (Active Comparator): Use of milk product with whey protein hydrolysate and Lacticaseibacillus rhamnosus GG
  Interventions: Dietary Supplement: Postbiotic and whey protein hydrolysate milk product

INTERVENTIONS:
Dietary Supplement: Placebo Comparator — Low-protein milk product
  Arms: Placebo milk product
Dietary Supplement: Whey protein hydrolysate milk product — Milk product with whey protein hydrolysate
  Arms: Whey protein hydrolysate milk product
Dietary Supplement: Postbiotic and whey protein hydrolysate milk product — Milk product with whey protein hydrolysate and Lacticaseibacillus rhamnosus GG
  Arms: Postbiotic and whey protein hydrolysate milk product

SUMMARY:
The aim of this intervention study is to investigate the effect of a specific postbiotic (Lacticaseibacillus rhamnosus GG = LGG) and whey protein on immunity, recovery, and weight management in young adults. The objective is based on previous knowledge about the health-promoting effects of these factors. A new goal is to study the combined effect of the postbiotic and whey protein. The results of the study can be utilized to promote the health of the young adults.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, 3-arm intervention involving young adults (n=160). Participants are randomized into three groups to receive different study product, and differences among the groups will be compared, for example, in terms of gut microbiota, weight changes, and inflammatory markers derived from blood samples.

ELIGIBILITY:
Inclusion Criteria:

- healthy

Exclusion Criteria:

* medicines and diseases that significantly affect the functioning of the stomach and intestines (e.g. irritable bowel syndrome)
* antibiotic treatment within 3 months
* asthma medication
* milk allergy (protein); the study product is lactose-free
* the participant must adhere to avoid the use of foods or nutritional supplements containing probiotics, and high-protein products, e.g. whey protein powders and high-protein snack bars

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Concentrations of inflammatory markers from the blood samples | At the baseline (week 0) and after eight weeks (last visit)
  hs-CRP (High-Sensitivity C-Reactive Protein), haptoglobin, suPAR (soluble urokinase-type Plasminogen Activator Receptor)

SECONDARY OUTCOMES:
Changes in the gut microbiota composition, diversity and function | At the baseline (week 0) and after eight weeks (last visit)
  Gut microbiota composition and function in feces by metagenomics shotgun sequencing
Weight of the participant | At the baseline (week 0), at four weeks and after eight weeks (last visit)
  Weight
Waist circumference of the participant | At the baseline (week 0) and after eight weeks (last visit)
  Waist circumference
Infections during the intervention | During intervention (Eight weeks)
  Self-reported infections during the intervention
Development of physical fitness | At the baseline (week 0) and after eight weeks (last visit)
  Based on walking test
Changes in the sleep quality | During intervention (Eight weeks)
  Monitoring sleep quality using a sports watch.
Changes in recovery | During intervention (Eight weeks)
  Monitoring recovery using a sports watch.
Blood pressure | At the baseline (week 0), at four weeks and after eight weeks (last visit)
  Blood pressure
BMI | At the baseline (week 0), at four weeks and after eight weeks (last visit)
  Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Laitinen, Professor, Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No